CLINICAL TRIAL: NCT02215512
Title: A Phase 1 Dose-Escalation Study of RRx-001 in Combination With Whole Brain Radiation in Subjects With Brain Metastases (BRAINSTORM)
Brief Title: Dose-Escalation Study of RRx-001 in Combination With Whole Brain Radiation in Subjects With Brain Metastases
Acronym: BRAINSTORM
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: EpicentRx, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: RRx001-22-01
Record Dates: First submitted 2014-08-11; First posted 2014-08-13 (Estimated); Last update posted 2021-11-03 (Actual); Status verified 2021-11

CONDITIONS: Brain Metastases
MeSH Terms: conditions — Brain Neoplasms | interventions — RRx-001

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- RRx-001 + WBRT (Experimental): RRx-001 administered intravenously twice a week (10, 17, 33, 55 mg) in subjects with brain metastases receiving whole brain radiation therapy (WBRT).
  Interventions: Drug: RRx-001 + WBRT

INTERVENTIONS:
Drug: RRx-001 + WBRT — Subjects will receive a combination of RRx-001 and whole brain radiotherapy.
  Other Names: Whole brain radiotherapy and RRx-001

SUMMARY:
In this dose-escalation study, the safety and tolerability of escalating dose levels of RRx-001 administered intravenously twice a week in subjects with brain metastases receiving whole brain radiation therapy (WBRT) will be assessed. Once a maximum tolerated dose is identified, further (up to approximately 30) participants will be recruited. The study will use MRI to monitor changes in tumor blood flow associated with RRx-001.

DETAILED DESCRIPTION:
The purpose of this research study is to test the safety and activity of whole brain radiation therapy with RRx-001, an experimental radiation sensitizer, in participants with brain metastases. As a radiation sensitizer, RRx-001 may increase the effect of whole brain radiation, the standard of care for brain metastases, on cancer cells in a specific target area while reducing damage to normal healthy cells. The ability to sensitize the cancer cells to radiation sets off a 'domino effect' of free radical damage in the tumor from a given amount or dose of radiation.

This study, which is called BRAINSTORM, since RRx-001 is associated with the development of a "free radical storm" in the brain tumors, is divided into two stages. In the first stage, approximately 3 participants at a time will be entered at a particular dose level of RRx-001 and then observed in order to see whether that dose results in side effects with radiation. If no bad side effects are observed, a second group of approximately 3 subjects will be given a slightly higher dose of RRx-001 and also monitored for side effects with radiation. This process will be repeated until a dose is reached, which has the most activity against the cancer cells without unacceptable side effects. At this point, more participants will be entered at this dose level until a maximum enrollment of approximately 30 participants has been reached.

RRx-001 releases a gas called nitric oxide, which widens the diameter of blood vessels, and allows the delivery of more oxygen to tumors. The presence of oxygen in tumors is critical for the effectiveness of radiation therapy, since cancer cells are about two to three times more vulnerable to radiation when oxygen is present. The reason that cancer cells are so much more vulnerable to the effects of radiation when oxygen is present is that radiation relies on the formation of harmful molecules known as free radicals that damage proteins and genetic material (DNA); without oxygen lower levels of free radicals are produced. Changes in the diameter go blood vessels will be studied by magnetic resonance imaging.

Unlike chemotherapies or other radiation sensitizers, RRx-001 does not have to enter the tumor to be effective because nitric oxide, as a gas, is able to spread or diffuse from the bloodstream into cancer cells.

ELIGIBILITY:
Inclusion Criteria:

* Written informed consent
* Age ≥18 years
* Eastern Cooperative Oncology Group (ECOG) performance status 0-2
* One or more brain metastases
* Prior radiation therapy to the brain is allowed with the exception of whole brain irradiation
* Subjects must be neurologically stable for at least 14 days prior to first dose of study drug;
* Male and female subjects who are not surgically sterile or post-menopausal must agree to use reliable methods of birth control for the duration of the study and for 90 days after the last dose of study drug administration; male partners of female subjects should use condoms for the duration of the study, and for 90 days after the last dose of study drug administration

Exclusion Criteria:

* Pregnant or lactating females
* Any evidence of severe or uncontrolled diseases
* Inadequate bone marrow reserve
* Previous whole brain radiotherapy
* Prior RRx-001 therapy
* Insufficient recovery from all side effects of previous anticancer therapies
* Evidence of blood clotting or bleeding abnormalities

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 29 (Actual)
Dates: Start 2015-02-06 (Actual); Primary Completion 2016-11-28 (Actual); Study Completion 2020-11-12 (Actual)

PRIMARY OUTCOMES:
Number, frequency and type of adverse events | 42 days
  To identify the maximum tolerated dose (MTD) of RRx-001 in combination with WBRT, defined as the dose of RRx-001 associated with a 20% probability of dose-limiting toxicity (DLT) in subjects with brain metastases

SECONDARY OUTCOMES:
Objective Response Rate | 4 months
  To assess the Objective Response Rate of RRx-001 in combination with WBRT using modified Response Evaluation Criteria in Solid Tumors
Clinical Benefit Rate | 4 months
  To assess the Clinical Benefit Rate of RRx-001 in combination with WBRT using modified Response Evaluation Criteria in Solid Tumors
Intracranial Progression Free Survival | 4 months
  To obtain a preliminary estimate of the efficacy of RRx-001 in combination with WBRT in prolonging intracranial Progression Free Survival in subjects with brain metastases
Overall Survival | 10 months
  Overall Survival in subjects with brain metastases treated with WBRT and RRx-001
Brain Imaging Parameters | 6 weeks
  To evaluate changes in imaging parameters of the brain as a surrogate measure of pharmacologic activity and neurocognitive outcome

CONTACTS AND LOCATIONS:
Overall Officials: Michelle Kim, MD, Principal Investigator — University of Michigan
Locations (5):
- United States (5):
  - Providence Saint John's Health Center, Santa Monica, California
  - University of Michigan, Ann Arbor, Michigan
  - Allegiance Health, Jackson, Michigan
  - Washington University School of Medicine, St Louis, Missouri
  - The Cancer Institute of New Jersey (Rutgers University), New Brunswick, New Jersey